CLINICAL TRIAL: NCT01825746
Title: My Own Health Report (MOHR): A Pragmatic Evaluation to Enhance Primary Care Based Goal Setting and Evidence-Based Support for Health Behavior and Psychosocial Issues Through Meaningful Use of Patient-Centered Data and Tools
Brief Title: Goal Setting for Health Behavior and Psychosocial Issues in Primary Care
Acronym: MOHR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Office of Behavioral and Social Sciences Research (OBSSR) (NIH); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VCUFM0001; U58DP002759-01 (NIH); R01CA140959 (NIH)
Record Dates: First submitted 2013-02-15; First posted 2013-04-08 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Health Behaviors; Obesity; Substance Abuse; Anxiety; Depression
MeSH Terms: conditions — Health Behavior; Obesity; Substance-Related Disorders; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early implementation practices (Active Comparator): 9 practices that will initially field the MOHR assessment for up to 6 months. These practices will serve as "intervention" sites for the effectiveness outcomes measured by the patient experience survey.
  Interventions: Other: Implementation of the MOHR assessment in primary care workflow
- Delayed implementation practices (Other): 9 practices that will field the MOHR assessment for up to 6 months but starting 4 months after the early implementation practices. These practices will serve as "control" sites for the effectiveness outcomes measured by the patient experience survey. However, they will provide intervention data with respect to Reach and cost during the delayed phase.
  Interventions: Other: Implementation of the MOHR assessment in primary care workflow

INTERVENTIONS:
Other: Implementation of the MOHR assessment in primary care workflow — The MOHR assessment includes (1) asking patients to complete the MOHR assessment on the web prior to encounters (available at www.MyOwnHealthReport.org it addresses10 distinct health behaviors and psychosocial issues including physical activity, diet, alcohol consumption, tobacco use, drug use, sleep, stress, depression and anxiety), (2) provision, via the tool, immediate patient feedback that includes identification of unhealthy issues, assessment of readiness to change, prioritization of issues to change, and preparation for goal-setting and action planning, (3) feedback to the primary care team on the patient status and priorities for change, (4) provision of counseling, goal setting, and referrals to local resources by clinicians during the subsequent office visit, and (5) follow-up with the clinicians and local resources as agreed upon by the patient and clinician.

SUMMARY:
The purpose of this delayed cluster randomized intervention trial is to evaluate primary care strategies to increase goal setting, shared decision-making and evidence-based support and counseling for health behaviors and psychosocial issues through the implementation of a standard set of practical, patient-centered survey items and related decision support tools, called the My Own Health Report (MOHR) assessment. Nine pairs of diverse primary care practices will participate, four pairs of federally qualified health centers clinics and 5 pairs of practice based research network practices. Practice pairs are similar in size, patient and staff mix, culture, and level of EHR integration. Within pairs, practices will be randomized to early or delayed intervention (4 months later). The intervention consists of implementing the MOHR assessment and patient counseling into clinical care for all patients presenting for wellness or chronic care during a 6 month study period. Prior to implementation, practices will receive brief training about health behavior counseling, goal setting, and action planning. Practices will also be provided materials to support evidence-based counseling and referrals to local community resources. MOHR assessment implementation details will be determined by each practice pair but will generally include (1) asking patients to complete the MOHR assessment on the web prior to encounters (available at www.MyOwnHealthReport.org it addresses10 distinct health behaviors and psychosocial issues including physical activity, diet, alcohol consumption, tobacco use, drug use, sleep, stress, depression and anxiety), (2) provision, via the tool, immediate patient feedback that includes identification of unhealthy issues, assessment of readiness to change, prioritization of issues to change, and preparation for goal-setting and action planning, (3) feedback to the primary care team on the patient status and priorities for change, (4) provision of counseling, goal setting, and referrals to local resources by clinicians during the subsequent office visit, and (5) follow-up with the clinicians and local resources as agreed upon by the patient and clinician. Data sources will include patient responses to the MOHR assessment, practice appointment records, and a patient experience survey mailed to the first 300 patients offered the MOHR assessment two weeks after their office visit. Primary outcomes will include the Reach and Effectiveness of the intervention. Reach will be assessed in early and delayed intervention sites when they field the MOHR assessment. Effectiveness will compare early and delayed intervention sites during the early intervention phase, allowing the delayed intervention sites to serve as controls. Reach outcomes will include the percent of eligible patients receiving and completing the MOHR assessment. Effectiveness outcomes will include the percent of patients reporting that they were asked about health topics, set a change goal, received assistance for making a change, were referred for local counseling and support, and/or made any changes. Additional outcomes will include maintenance of the MOHR assessment implementation beyond 4 months, changes in patient reported health behavior and psychosocial measures by repeated administration of the MOHR assessment 4 months after initial completion, qualitative assessments on implementation factors and context that influence outcomes, and cost, in terms of time and resources required for practices to implement the MOHR assessment.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients presenting for chronic or wellness care at the study practices

Exclusion Criteria:

* Acute illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3591 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Reach | Entire 6 month early or delayed implementation phase
  The percent of eligible patients (e.g. those presenting for wellness or chronic care) who are offered the MOHR assessment and who complete the MOHR assessment
Effectiveness - Ask | 6 month early implementation phase
  The percent of patients reporting that they were asked about health behavior and psychosocial topics in the early implementation (intervention) versus the delayed implementation (control) practices
Effectiveness - Goal Setting | 6 month early implementation phase
  The percent of patients reporting that they set a goal about health behavior and psychosocial topics in the early implementation (intervention) versus the delayed implementation (control) practices
Effectiveness - Assistance | 6 month early implementation phase
  The percent of patients reporting that received assistance for health behavior and psychosocial topic in the early implementation (intervention) versus the delayed implementation (control) practices
Effectiveness - Referred | 6 month early implementation phase
  The percent of patients reporting that they were referred for health behavior and psychosocial counseling to a local program in the early implementation (intervention) versus the delayed implementation (control) practices

SECONDARY OUTCOMES:
Cost | 6 month early and delayed implementation phase
  The cost in terms of resources and time for practice to implement and field the MOHR assessment
Health behavior and psychosocial changes | 4 months after completion of the initial MOHR assessment
  The change in patient responses to the 10 health behavior and psychosocial domains of the MOHR assessment with re-administration 4 months after initial completion

CONTACTS AND LOCATIONS:
Overall Officials: Alex H Krist, MD MPH, Principal Investigator — Virginia Commonwealth University
Locations (8):
- United States (8):
  - UCLA Fielding School of Public Health, Los Angeles, California
  - University of North Carolina, Chapel Hill, North Carolina
  - OCHIN, Portland, Oregon
  - Department of Health Promotion and Community Health Sciences, Texas A&M Health Sciences Center School of Rural Public Health, College Station, Texas
  - University of Texas School of Public Health, Houston, Texas
  - Vermont College of Medicine, Burlington, Vermont
  - Virginia Ambulatory Care Outcomes Research Network, Richmond, Virginia
  - Carilion Health System, Roanoke, Virginia

REFERENCES:
- [Background] Estabrooks PA, Boyle M, Emmons KM, Glasgow RE, Hesse BW, Kaplan RM, Krist AH, Moser RP, Taylor MV. Harmonized patient-reported data elements in the electronic health record: supporting meaningful use by primary care action on health behaviors and key psychosocial factors. J Am Med Inform Assoc. 2012 Jul-Aug;19(4):575-82. doi: 10.1136/amiajnl-2011-000576. Epub 2012 Apr 17. PMID 22511015
- [Derived] Krist AH, Glasgow RE, Heurtin-Roberts S, Sabo RT, Roby DH, Gorin SN, Balasubramanian BA, Estabrooks PA, Ory MG, Glenn BA, Phillips SM, Kessler R, Johnson SB, Rohweder CL, Fernandez ME; MOHR Study Group. The impact of behavioral and mental health risk assessments on goal setting in primary care. Transl Behav Med. 2016 Jun;6(2):212-9. doi: 10.1007/s13142-015-0384-2. PMID 27356991
- [Derived] Krist AH, Phillips SM, Sabo RT, Balasubramanian BA, Heurtin-Roberts S, Ory MG, Johnson SB, Sheinfeld-Gorin SN, Estabrooks PA, Ritzwoller DP, Glasgow RE; MOHR Study Group. Adoption, reach, implementation, and maintenance of a behavioral and mental health assessment in primary care. Ann Fam Med. 2014 Nov-Dec;12(6):525-33. doi: 10.1370/afm.1710. PMID 25384814
- [Derived] Phillips SM, Glasgow RE, Bello G, Ory MG, Glenn BA, Sheinfeld-Gorin SN, Sabo RT, Heurtin-Roberts S, Johnson SB, Krist AH; MOHR Study Group. Frequency and prioritization of patient health risks from a structured health risk assessment. Ann Fam Med. 2014 Nov-Dec;12(6):505-13. doi: 10.1370/afm.1717. PMID 25384812
- [Derived] Krist AH, Glenn BA, Glasgow RE, Balasubramanian BA, Chambers DA, Fernandez ME, Heurtin-Roberts S, Kessler R, Ory MG, Phillips SM, Ritzwoller DP, Roby DH, Rodriguez HP, Sabo RT, Sheinfeld Gorin SN, Stange KC; MOHR Study Group. Designing a valid randomized pragmatic primary care implementation trial: the my own health report (MOHR) project. Implement Sci. 2013 Jun 25;8:73. doi: 10.1186/1748-5908-8-73. PMID 23799943
- See also: Grid Enabled Measures Database used to help collect health behavior and psychosocial measures to consider for inclusion on the MOHR assessment — https://www.gem-beta.org